CLINICAL TRIAL: NCT05751278
Title: A Randomized Trial of Cryoprobe Versus Forceps for Transbronchial Biopsy
Brief Title: Cryoprobe Versus Forceps for Transbronchial Biopsy
Acronym: FROSTBITE-2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Erbe USA Incorporated (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: IRB00344800
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Lung Diseases
Keywords: lung; cryoprobe; bronchoscopic; biopsy
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Cryoprobe (Experimental): Participants in this arm will undergo a standard of care bronchoscopy with a transbronchial biopsy using the 1.1mm sheath cryoprobe
  Interventions: Device: ERBECRYO® 2 Cryosurgical Unit and Accessories - K190651
- Forceps (Active Comparator): Participants in this arm will undergo a standard of care bronchoscopy with a transbronchial biopsy using forceps
  Interventions: Device: Radial Jaw 4 Pulmonary Biopsy Forceps

INTERVENTIONS:
Device: ERBECRYO® 2 Cryosurgical Unit and Accessories - K190651 — ERBE 1.1mm flexible single-use cryoprobe with oversheath
  Arms: Cryoprobe
Device: Radial Jaw 4 Pulmonary Biopsy Forceps — Radial Jaw 4 Pulmonary Biopsy Forceps Standard Capacity for 2mm endoscope
  Arms: Forceps

SUMMARY:
The purpose of this study is to compare the effectiveness of transbronchial biopsy done by a 1.1mm cryoprobe versus the standard 2.0mm forceps.

DETAILED DESCRIPTION:
A smaller (1.1mm), flexible, single-use cryoprobe with an oversheath has been developed that can be used for transbronchial biopsies. This device has the potential to gather larger and higher quality tissue samples than the standard method using forceps, and with potentially fewer complications than older, larger versions of the cryoprobe.

For this study, patients will be randomized in a 1:1 fashion to transbronchial biopsy using a 1.1 mm cryoprobe versus 2.0 mm forceps, stratified by indication (evaluation of lung transplant allograft, diffuse parenchymal lung disease or pulmonary parenchymal lesion). Blinding of the proceduralist is not possible due to the nature of the procedure. Pathologists interpreting the biopsy samples will be blinded to the biopsy device used.

Patients enrolled in this study will have data collected by research staff for up to 30 days after the bronchoscopic biopsy procedure is performed. This 30-day follow-up period is the standard of care following bronchoscopic biopsy procedures.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, ≥ 18-years-old
* Scheduled to undergo bronchoscopy with transbronchial biopsy per standard of care

Exclusion Criteria:

* Pregnant or nursing woman or woman of child-bearing potential who refuse to take a pregnancy test prior to enrollment
* Severe pulmonary hypertension (RVSP > 60 mmHg)
* Stroke within the last 6 months or myocardial infarction within the last 3 months
* Presence of bleeding disorder
* Platelet count < 50,000 per mL at time of enrollment
* Use of systemic anticoagulation or antiplatelet therapy without the ability to hold therapy for the recommended time prior to invasive procedure (aspirin monotherapy is acceptable)
* Do Not Resuscitate (DNR) status
* Do Not Intubate (DNI) status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield as assessed by number of patients for which the procedure led to a diagnosis | During procedure, up to 1 hour
  Diagnostic Yield as Assessed by Number of Patients for Which the Procedure [Cryobiopsy or Forceps] Led to a Diagnosis.

SECONDARY OUTCOMES:
Diagnostic yield for pulmonary parenchymal lesions | During procedure, up to 1 hour
  Diagnostic Yield as Assessed by Number of Patients with pulmonary parenchymal lesions for Which the Procedure [Cryobiopsy or Forceps] Led to a Diagnosis.
Diagnostic yield for diffuse parenchymal lung disease | During procedure, up to 1 hour
  Diagnostic Yield as Assessed by Number of Patients with diffuse parenchymal lung disease for Which the Procedure [Cryobiopsy or Forceps] Led to a Diagnosis.
Diagnostic yield for Lung Transplant | During procedure, up to 1 hour
  Diagnostic Yield as Assessed by Number of Patients with a Lung Transplant for Which the Procedure [Cryobiopsy or Forceps] Led to a Diagnosis.
Histological Accessibility grade of the biopsy specimen | Participants assessed for the outcome measure at the time of biopsy procedure (up to 1 hour)
  7-point Likert scale: 0-6 with 0 being worse and 6 being best.
Bleeding Complication Rate | Within 30 days of procedure
  Number of occurrences of bleeding (grade ≥ 3 modified CTCAE).
Pneumothorax Complication Rate | Within 30 days of procedure
  Number of occurrences of pneumothorax requiring chest tube placement (grade ≥ 2, CTCAE).
Post-Procedure Respiratory Failure Rate | Within 30 days of procedure
  Number of occurrences of post-procedure respiratory failure (defined as the need for non-invasive or mechanical ventilation requiring ICU admission).
Number of deaths | Within 30 days of procedure
  Number of occurrences of death.
Total Histologic Area | Participants assessed for the outcome measure at the time of biopsy procedure (up to 1 hour)
  Total Histologic Area in Square Millimeters.
Alveolated Area | Participants assessed for the outcome measure at the time of biopsy procedure (up to 1 hour)
  Alveolated Area Square Millimeters
Percent Crush Artifact | Participants assessed for the outcome measure at the time of biopsy procedure (up to 1 hour)
  Percent total area for Crush Artifact.
Artifact-free lung parenchyma | Participants assessed for the outcome measure at the time of biopsy procedure (up to 1 hour)
  Percent Artifact-free lung parenchyma.
Adequacy for Molecular Testing | Participants assessed for the outcome measure at the time of biopsy procedure (up to 1 hour)
  Assessed as a yes or no using Next Generation Sequencing (NGS).
Activation Time | At the time of procedure, up to 1 hour
  Activation Time in Seconds.
Procedure Time | At the time of procedure, up to 1 hour
  Procedure Time Seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Thiboutot, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (7):
- United States (7):
  - Northwestern Medicine, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - NYU Langone Health, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - The Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center (VUMC), Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No